CLINICAL TRIAL: NCT03859076
Title: Mindfulness Based Blood Pressure Reduction: Stage 2a Randomized Controlled Trial
Brief Title: UH3 Phase - Mindfulness-Based Blood Pressure Reduction (MB-BP) : Stage 2a RCT
Acronym: MB-BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1412001171-2; 5UH3AT009145-04 (NIH)
Record Dates: First submitted 2019-02-20; First posted 2019-03-01 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Hypertension; Prehypertension
Keywords: mindfulness; blood pressure; hypertension; prehypertension; self regulation; Science of Behavior Change; attention control; self awareness; emotion regulation
MeSH Terms: conditions — Hypertension; Prehypertension; Self-Control; Emotional Regulation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will implement blinding of staff performing participant assessments and data analysts performing statistical analyses. The principal investigator will be blinded to group allocation, except for participants that he is involved with instructing in the MB-BP intervention (there are multiple instructors). The prinicipal investigator has no access to the master data file. Equipoise is emphasized for all staff who interact with participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MB-BP Intervention (Experimental): MB-BP customizes Mindfulness-Based Stress Reduction (MBSR) to participants with hypertension. It consists of nine 2.5-hour weekly group sessions & a 7.5-hour one-day session. Content includes education on hypertension risk factors, hypertension health effects, & specific mindfulness modules focused on awareness of BP determinants such as diet, physical activity, anti-hypertensive medication adherence, alcohol consumption, & stress reactivity. Students learn a range of mindfulness skills (body scan exercises, meditation and yoga). Participants are given a home BP monitor. Participants with uncontrolled hypertension are offered to have their physicians notified; for those without a physician, the investigator works to provide access within health insurance constraints.
  Interventions: Behavioral: MB-BP
- Enhanced Usual Care Control (Active Comparator): Those in the control group receive an educational brochure from the American Heart Association (product code 50-1731) and a validated home blood pressure monitor (Omron, Model PB786N), that has an evidence-based approach to lower blood pressure. All participants who have uncontrolled hypertension (blood pressure >140/90 mmHg) will be offered to have their physicians notified, if not already being overseen for it. For participants with uncontrolled hypertension who do not have a physician, the investigator works to provide access within constraints of their health insurance. Additionally, participants randomized to the control group are asked to refrain from engaging in any type of formal mindfulness practice more than weekly during the first six months of study involvement.
  Interventions: Other: Enhanced Usual Care Control

INTERVENTIONS:
Behavioral: MB-BP — MB-BP customizes Mindfulness-Based Stress Reduction (MBSR) to participants with hypertension. It consists of nine 2.5-hour weekly group sessions & a 7.5-hour one-day session. Content includes education on hypertension risk factors, hypertension health effects, & specific mindfulness modules focused on awareness of BP determinants such as diet, physical activity, anti-hypertensive medication adherence, alcohol consumption, & stress reactivity. Students learn a range of mindfulness skills (body scan exercises, meditation and yoga). Participants are given a home BP monitor. Participants with uncontrolled hypertension are offered to have their physicians notified; for those without a physician, the investigator works to provide access within health insurance constraints.
  Arms: MB-BP Intervention
Other: Enhanced Usual Care Control — Those in the control group receive an educational brochure from the American Heart Association (product code 50-1731) and a validated home blood pressure monitor (Omron, Model PB786N), that has an evidence-based approach to lower blood pressure. All participants who have uncontrolled hypertension (blood pressure >140/90 mmHg) will be offered to have their physicians notified, if not already being overseen for it. For participants with uncontrolled hypertension who do not have a physician, the investigator works to provide access within constraints of their health insurance. Additionally, participants randomized to the control group are asked to refrain from engaging in any type of formal mindfulness practice more than weekly during the first six months of study involvement.
  Arms: Enhanced Usual Care Control

SUMMARY:
The primary aim is to identify the impacts of a behavioral intervention called "Mindfulness-Based Blood Pressure Reduction" (MB-BP) vs. enhanced usual care on the primary self-regulation target, specifically an assay of self-related processes (Multidimensional Assessment of Interoceptive Awareness) (MAIA) at 6 months, via a randomized controlled trial.

DETAILED DESCRIPTION:
Effects of mindfulness interventions customized for prehypertensive/hypertensive patients are poorly understood. Until methodologically rigorous studies to evaluate customized interventions for hypertension are performed, it will be unknown whether the observed preliminary effects of general mindfulness interventions on blood pressure reduction could be much more effective with a tailored approach. Consequently, this study proposes to conduct a behavioral intervention study to evaluate whether Mindfulness-Based Stress Reduction (MBSR) customized to prehypertensive and hypertensive patients has the potential to provide clinically relevant reductions in blood pressure.

This customized intervention is called Mindfulness-Based Blood Pressure Reduction (MB-BP). The study follows the NIH Stage Model for Behavioral Intervention Development, where targets likely proximally affected by the intervention are identified, that should also have effect on the longer-term outcomes (e.g. blood pressure, mortality). The selected targets, consistent with theoretical frameworks and early evidence how mindfulness interventions could influence mental and physical health outcomes, are measures of self-regulation including (1) attention control (specifically the Sustained Attention Response Task and Mindful Attention Awareness Scale), (2) emotion regulation (specifically the Pittsburgh Stress Battery and the Perceived Stress Scale), and (3) self-awareness (specifically the Heart Beat Detection Task and Multidimensional Assessment of Interoceptive Awareness). Based on the degree of target engagement, MB-BP can be further customized to better engage with the targets as needed.

ELIGIBILITY:
Inclusion Criteria:

* Elevated blood pressure or hypertension defined as ≥120 mmHg systolic or ≥80 mmHg diastolic pressure.
* Able to speak, read, and write in English.
* All adults (≥18 years of age), genders and racial/ethnic groups are eligible to be included.

Exclusion Criteria:

Exclusion criteria follow standard guidelines and recommendations:

* current regular mindfulness meditation practice (>once/week)
* serious medical illness or cognitive condition (e.g., dementia) precluding regular class attendance and/or participation
* current substance abuse, suicidal ideation or eating disorder
* history of bipolar or psychotic disorders or self-injurious behaviors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Self-Regulation Primary Outcome: Multidimensional Assessment of Interoceptive Awareness (MAIA) | 6 month follow-up
  a validated measure of body awareness - a 32 item self-report measure composed of the following 8 subscales: (i) Noticing, (ii) Not-Distracting, (iii) Not-Worrying, (iv) Attention Regulation, (v) Emotional Awareness, (vi) Self-Regulation, (vii) Body Listening, and (viii) Trusting. Individuals rate items using a 6 point Likert scale from 0 ('Never') to 5 ('Always'). Total scores are obtained through reverse coding items 5, 6, 7, 8, 9 and summing all items. Higher scores indicate higher levels of positive awareness.

SECONDARY OUTCOMES:
Heartbeat Detection Task | Baseline, 10 weeks, 6 months
  Behavioral measure of self-awareness
Interoceptive Awareness fMRI Task | Baseline, 10-week follow-up
  Those who elect to take part in the fMRI study will undergo an fMRI scanning session for approximately 40 minutes. Scans will be acquired with a 3T scanner while the subject is in the resting state. Participants will undergo a separate informed consent and screening process for the fMRI imaging, so that they can be in the MB-BP study without imaging if they prefer.
Difficulties in Emotion Regulation Scale (DERS) | Baseline, 10 weeks, 6 months
  Behavioral measure of emotion regulation - The Difficulties in Emotion Regulation Scale is a 36-item self-report measure of six facets of emotion regulation. Items are rated on a scale of 1-5, with 1 being ("almost never [0-10%]"); 2 ("sometimes [11-35%]"); 3 ("about half the time [36-65%]"); 4 ("most of the time [66-90%]); and 5 being ("almost always [91-100%]"). Higher scores indicate more difficulty in emotion regulation.
Pittsburgh Stress Battery | Baseline, 10 weeks, 6 months
  Behavioral measure of stress reactivity
Perceived Stress Scale (PSS-14) | Baseline, 10 weeks, 6 months
  14-item self-report measure of perceived stress - Participants indicate how often they have found their lives unpredictable, uncontrollable, and overloaded in the last month. Items are rated on a 4 point Likert scale with 0 being ("Never"); 1 ("Almost Never"); 2 ("Sometimes"); 3 ("Fairly often") and 4 ("Very often"). PSS-14 scores are obtained by reversing the scores on the seven positive items, e.g., 0=4, 1=3, 2=2, etc., and then summing across all 14 items. Items 4, 5, 6, 7, 9, 10, and 13 are the positively stated items.
Anxiety Symptoms - self-report | Baseline, 10 weeks, 6 months
  Assessed via the Beck Anxiety Inventory (BAI) scale. The BAI is a 21-item self-report measure of anxiety. Participants indicate how much they have been bothered by an anxiety symptom during the past month. Items are rated on a 3-point Likert scale with 0 being "Never"); 2 ("Mildly but it didn't bother me much"); 2 ("Moderately - it wasn't pleasant at times"); 3 ("Severely- it bothered me a lot"). The total score is calculated by finding the sum of the 21 items. A score of 0-21= low anxiety, Score of 22-35 = moderate anxiety, Score of 36 and above = potentially concerning levels of anxiety.
Depressive Symptoms - self-report | Baseline, 10 weeks, 6 months
  Assessed via Center for Epidemiologic Studies Depression Scale Revised (CESD-R). The CESD-R is a 20-item self-report measure of depression in nine different groups according to the DSM-5. The symptom groups are Sadness (items 2,4,6), Loss of Interest (items 8, 10), Appetite (1,18), Sleep (5,11,19), Thinking/Concentration (3,20), Guilt (9,17), Tired (7,16), Movement (12,13), and Suicidal Ideation (14,15). Response values for each question are 0 ("Not at all or less than one day"); 1 ("1-2 days"); 2 ("3-4 days); 3 ("5-7 days"); 4 ("Nearly every day for 2 weeks"). The total score is calculated as a sum of responses to all 20 questions.
Sustained Attention to Response Task (SART) | 6 month follow-up
  Behavioral measure of attention control - The Sustained Attention to Response Task (SART) is a computer-based go/no-go task that requires participants to withhold behavioral response to a single, infrequent target (often the digit 3) presented amongst a background of frequent non-targets (0-2, 4-9). After each block, two probe questions are presented in succession. The first asks, "Where was your attention focused during this block of trials?" Participants respond on a 6-point Likert scale, where 1 represents, "on task, " and 6, "off task." A second question asks, "How aware were you of where your attention was during this block of trials?" Participants respond on a similar scale, where 1 represents, "aware, " and 6, "unaware."
Self-Compassion | 6 months
  Assessed using the 12-item validated Self-Compassion Scale Short Form (SCS-SF); Participants indicate how they typically act towards themselves in difficult times using a 5-point Likert scale with 1 being "Almost Never" to 5 being "Almost Always". The total self-compassion score is calculated by reverse scoring the negative subscale items -self-judgment, isolation, and over-identification (i.e., 1 = 5, 2 = 4, 3 = 3, 4 = 2, 5 = 1) then computing a total mean.
Self-Efficacy | Baseline, 10 weeks, 6 months
  Assessed using the validated Self-Control Scale short form and the SECD-6 Scale. The Self Control Scale measures self-control. The scale consists of 36 items, measured on a scale from 1, "not at all like me" to 5, "very much like me."
Dietary Approaches to Stop Hypertension (DASH)-consistent diet | 6 month follow-up
  Self-report via Willet Food Frequency Questionnaire. Participants are asked to fill in the circle indicating how often on average they have used the food item during the past year. Response categories include "Never, or less than once per month", "1-3 per month"; "1 per week"; "2-4 per week"; "5-6 per week"; "1 per day"; "2-3 per day"; "4-5 per day"; "6+ per day."
Alcohol consumption - self report | 6 month-follow up
  Self-report via Willet Food Frequency Questionnaire. Participants are asked to fill in the circle indicating how often on average they have used the food item during the past year. Response categories include "Never, or less than once per month", "1-3 per month"; "1 per week"; "2-4 per week"; "5-6 per week"; "1 per day"; "2-3 per day"; "4-5 per day"; "6+ per day."
Electronically-Measured Antihypertensive Medication Adherence | 6 months
  Measured continuously using electronic medication bottle caps (eCAPS, Ottawa, Canada)
Body Mass Index | Baseline, 10 weeks, 6 months
  Height and weight directly assessed using standard epidemiologic methods, with change evaluated in participants considered overweight or obese (BMI≥25kg/m)
Physical Activity - self report | Baseline, 10 weeks, 6 months
  Assessed via the International Physical Activity Questionnaire (IPAQ). The IPAQ is a 27-item self-reported measure of physical activity. Duration (minutes) and frequency (days) of physical activity in the last seven days is measured in 5 domains (1: job related; 2: transportation; 3: housework, house maintenance, caring for family; 4: Recreation, sport, and leisure time; 5: Time spent sitting). Overall score is calculated using responses to all questions. Amount of physical activity places participant in 1 of 3 categories: 1) Low/inactive; 2) Moderate; 3) High.

CONTACTS AND LOCATIONS:
Overall Officials: Eric B Loucks, PhD, Principal Investigator — Brown University
Locations (1):
- Brown Mindfulness Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Loucks EB, Kronish IM, Saadeh FB, Scarpaci MM, Proulx JA, Gutman R, Britton WB, Schuman-Olivier Z. Adapted Mindfulness Training for Interoception and Adherence to the DASH Diet: A Phase 2 Randomized Clinical Trial. JAMA Netw Open. 2023 Nov 1;6(11):e2339243. doi: 10.1001/jamanetworkopen.2023.39243. PMID 37917063
- [Derived] Loucks EB, Kronish IM, Saadeh FB, Scarpaci MM, Proulx JA, Gutman R, Britton WB, Schuman-Olivier Z. Effects of Adapted Mindfulness Training on Interoception and Adherence to the Dietary Approaches to Stop Hypertension (DASH) Diet: The MB-BP Randomized Clinical Trial. medRxiv [Preprint]. 2023 May 15:2023.05.10.23289818. doi: 10.1101/2023.05.10.23289818. PMID 37292774
- [Derived] Loucks EB, Schuman-Olivier Z, Saadeh FB, Scarpaci MM, Nardi WR, Proulx JA, Gutman R, King J, Britton WB, Kronish IM. Effect of Adapted Mindfulness Training in Participants With Elevated Office Blood Pressure: The MB-BP Study: A Randomized Clinical Trial. J Am Heart Assoc. 2023 Jun 6;12(11):e028712. doi: 10.1161/JAHA.122.028712. Epub 2023 May 23. PMID 37218591

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT03859076/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT03859076/ICF_001.pdf